CLINICAL TRIAL: NCT05230550
Title: Post-Marketing Surveillance (Special Use-results Surveillance on Long-term Use) With Sogroya® A Multi-centre, Prospective, Open Label, Single-arm, Observational, Non-interventional Post-marketing Study to Investigate the Long-term Safety and Clinical Parameters of Sogroya® Therapy in Patients With Adult Growth Hormone Deficiency (AGHD) (Only Severe Case) Under Normal Clinical Practice Conditions in Japan
Brief Title: Post-Marketing Surveillance (Special Use-results Surveillance on Long-term Use) With Sogroya®
Status: Enrolling by invitation | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN8640-4638; U1111-1247-5417 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-01-28; First posted 2022-02-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Adult Growth Hormone Deficiency
MeSH Terms: conditions — Dwarfism, Pituitary | interventions — somapacitan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with AGHD (only severe case): Participants will be treated with commercially available Sogroya® according to routine clinical practice at the discretion of the treating physician. The decision to treat a patient with Sogroya® has been made at the treating physician's discretion and independently from the decision to include the patient in this study.
  Interventions: Drug: Somapacitan

INTERVENTIONS:
Drug: Somapacitan — Sogroya® therapy in participants with AGHD (only severe case) under normal clinical practice conditions
  Other Names: Sogroya®

SUMMARY:
Participants are invited to take part in this study because they have AGHD (only severe case). The purpose of this study is to assess long term safety and effectiveness of Sogroya® in patients with AGHD (only severe case) under normal clinical practice condition in Japan. Participants will get Sogroya® as prescribed by the study doctor. Participants will be in the study for about 2 to 5 years depending on when they take part in the study. Participants will be asked to fill in the quality of life questionnaires.

ELIGIBILITY:
Inclusion Criteria:

1. Signed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol)
2. The decision to initiate treatment with commercially available Sogroya® has been made by the patient/LAR and the treating physician before and independently from the decision to include the patient in this study.
3. Male or female, no age limitation
4. Diagnosis of AGHD (only severe case)
5. GH treatment naïve ("naïve patients") or "switched patients". "Naïve patients" are patients who are not exposed to any GH product to date or patients who were exposed to other GH product more than 180 days prior to registration. "Switched patients" are patients who is now treated by other GH product or patients who were exposed to other GH product within 180 days prior to registration.

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study
2. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
3. Patients with hypersensitivity to the active substance or to any of the excipients
4. Patients with malignant tumor
5. Female patients who are either pregnant or likely to be pregnant

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Adult Growth Hormone Deficiency (only severe case)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of adverse events | From baseline (week 0) to end of study (up to 260 weeks)
  Measured as number
Number of serious adverse events | From baseline (week 0) to end of study (up to 260 weeks)
  Measured as number
Number of serious adverse reactions | From baseline (week 0) to end of study (up to 260 weeks)
  Measured as number
Number of adverse reactions | From baseline (week 0) to end of study (up to 260 weeks)
  Measured as number

SECONDARY OUTCOMES:
Change in body fat mass | From baseline (week 0) to end of study (up to 260 weeks)
  Measured as kilogram (kg)
Change in body fat percentage | From baseline (week 0) to end of study (up to 260 weeks)
  Measured as percent (%)
Change in lean body mass | From baseline (week 0) to end of study (up to 260 weeks)
  Measured as kg
Change in cross-sectional total adipose tissue compartments (TAT) | From baseline (week 0) to end of study (up to 260 weeks)
  Measured as square centimeter (cm^2)
Change in subcutaneous adipose tissue compartments (SAT) | From baseline (week 0) to end of study (up to 260 weeks)
  Measured as cm^2
Change in visceral adipose tissue compartments (VAT) | From baseline (week 0) to end of study (up to 260 weeks)
  Measured as cm^2
Change in Total cholesterol (T-Cho) | From baseline (week 0) to end of study (up to 260 weeks)
  Measured as milligrams per deciliter (mg/dL)
Change in Low Density Lipoprotein-Cholesterol (LDL-Cho) | From baseline (week 0) to end of study (up to 260 weeks)
  Measured as mg/dL
Change in High Density Lipoprotein-Cholesterol (HDL-Cho) | From baseline (week 0) to end of study (up to 260 weeks)
  Measured as mg/dL
Change in triglyceride | From baseline (week 0) to end of study (up to 260 weeks)
  Measured as mg/dL
Change in Insulin-like Growth Factor I (IGF-I) standard deviation score (SDS) | From baseline (week 0) to end of study (up to 260 weeks)
  Measured as standard deviation score
Change in Quality of Life (QOL) Adult Hypopituitarism Questionnaire (AHQ) score | From baseline (week 0) to end of study (up to 260 weeks)
  Measured as score range (0 = unfavorable to 6 = favorable)
Change in QOL Treatment Related Impact Measure-Adult Growth Hormone Deficiency (TRIM-AGHD) score | From baseline (week 0) to end of study (up to 260 weeks)
  Measured as score range (1 to 5; lower score indicates a better health state)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency dept. 2834, Study Director — Novo Nordisk A/S
Locations (47):
- Japan (47):
  - Ikeda Hospital, Diabetes Medicine, Amagasaki-shi, Hyogo
  - University of Yamanashi Hospital, Chuo-shi, Yamanashi-ken
  - Fukuoka University Chikushi Hospital_Endocrinology and Diabetes Mellitus, Fukuoka
  - Kurume University Hospital, Fukuoka
  - Fukuoka University Hospital, Fukuoka-shi, Fukuoka-ken
  - Kyushu University Hospital, Fukuoka-shi, Fukuoka
  - Gifu University Hospital, Gifu
  - Tsugaru General Hospital, Goshogawara-shi, Aomori-ken
  - Gunma University Hospital, Dept. of Endocrinology and Diabetes, Gunma
  - Hamamatsu University Hospital, Hamamatsu-shi, Shizuoka
  - Hirosaki University Hospital, Hirosaki-shi, Aomori-ken
  - Hyogo Prefectural Kakogawa Medical Center, Hyōgo
  - Takara Clinic, Iida-shi, Nagano-ken
  - Shimane Univ. HP, Dept of Endocrinology&Metabolism, Izumo, Shimane
  - Joetsu General Hospital, Joetsu-shi, Niigata-ken
  - Kagoshima Medical Center, Kagoshima-shi, Kagoshima-ken
  - Kagoshima University Hospital_Neurosurgery, Kagoshima-shi, Kagoshima
  - Yokohama Medical Center, Kanagawa
  - Kitasato University Hospital, Kanagawa
  - Nara Medical University Hospital_Kashihara-shi, Nara, Kashihara-shi, Nara
  - Nippon Medical School Musashikosugi Hospital_Neurological Surgery, Kawasaki-shi, Kanagawa
  - Kobe University Hospital, Kobe-shi, Hyogo
  - Konan Hospital, Kumamoto
  - Kumamoto University Hospital, Diabetes, Metabo and Endo, Kumamoto-shi, Kumamoto
  - Kyoto University Hospital, Kyoto-shi, Kyoto
  - Toranomon Hospital, Endocrinology and Metabolism, Minato-ku, Tokyo
  - University of Miyazaki Hospital, Miyazaki-shi, Miyazaki-ken
  - Aichi Medical University Hospital, Nagakute-shi, Aichi
  - Okamoto Internal Medicine and Pediatrics Clinic, Nara
  - Kurebayashi Diabetes Clinic, Nishinomiya-shi, Hyogo-ken
  - Okayama University Hospital_General Medicine, Okayama-shi, Okayama
  - Osaka Endocrine Clinic, Osaka
  - Kibounomori Clinic, Osaka
  - Osaka City University Hospital, Osaka
  - Yasuhara Children's Clinic, Osaka
  - Osaka Women's and Children's Hospital, Osaka
  - NTT East Japan Sapporo HP, Diabetes Mellitus & Int med Endo, Sapporo, Hokkaido
  - JCHO Sendai Hospital, Sendai-shi, Miyagi-ken
  - Omi Medical Center, Shiga
  - Hamamatsu-kita-Hospital, Shizuoka
  - Hamamatsu Medical Center, Shizuoka
  - Shizuoka General Hospital, Shizuoka-shi, Shizuoka-ken
  - Tochigi Medical Center Shimotsuga, Tochigi-shi, Tochigi-ken
  - Hosaka Kodomo Clinic, Tokyo
  - Ehime University Hospital, Toon-shi, Ehime
  - Tottori University Hospital_Endocrinology and Metabolism, Tottori
  - Yamagata University Hospital, Internal Medicine 3, Yamagata-shi, Yamagata

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com
URL: http://novonordisk-trials.com